CLINICAL TRIAL: NCT06155422
Title: Efficacy and Safety of Cadonilimab (PD-1/CTLA-4 Bispecific Antibody) in the Treatment of Recurrent or Metastatic Cervical Cancer: a Multicenter, Prospective, Real-world Study
Brief Title: A Prospective Real-world Study of Cadonilimab in Patients With Recurrent or Metastatic Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Gang Chen (101199) (Other)
Responsible Party: Sponsor-Investigator, Gang Chen (101199), Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: AK104-RWS-002
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-09

CONDITIONS: Recurrent or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cadonilimab-treated Recurrent or Metastatic Cervical Cancer
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — recurrent or metastatic cervical cancer in the first, second or third lines Systematic treatment

SUMMARY:
This real-world study included all patients with recurrent or metastatic cervical cancer who used Cadonilimab in clinical practice, regardless of treatment lines and combination with different treatments. Through follow-up observations, the aim of this study is to analyze the efficacy of Cadonilimab for recurrent or metastatic cervical cancer in the real world, and to explore the differences in the efficacy of Cadonilimab in different stages of treatment, as well as the efficacy of different treatment combinations, so as to provide clinical evidence for the use of Cadonilimab for recurrent or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form (ICF) voluntarily.
2. Aged ≥ 18years, female.
3. Histologically or cytologically confirmed cervical cancer, ① recurrent or metastatic (FIGO IVB) cervical cancer, not amenable to curative surgery or concurrent chemoradiotherapy, no prior systemic therapy for persistent, recurrent or metastatic disease, or ② subjects have demonstrated radiologically confirmed disease progression during or after last treatment, subjects will have no more than 2 lines of systemic therapy in the recurrence or metastatic stages. neoadjuvant chemotherapy, adjuvant chemotherapy, or Chemotherapy of non-recurrent or metastatic stage chemoradiotherapy,will not be counted as a treatment line number.
4. The histological types include squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma.
5. At least 1 measurable lesion per RECIST v1.1, which is applicable for repeated accurate measurement.
6. Life expectancy> 12 weeks.
7. Adequate organ function.
8. Female patients with fertility must have a urine or serum pregnancy test within 3 days before the first medication (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test is required, based on the serum pregnancy result), and the result is negative. If a fertile female patient has sex with an unsterilized male partner, the patient must use an acceptable contraceptive method since screening and must consent to continued use of the contraceptive method for 120 days after the last administration of the study drug; Whether to stop contraception after this time point should be discussed with the investigator
9. Subjects must be willing and able to comply with the scheduled visits, treatment regimens, laboratory tests, and other requirements in the study.

Exclusion Criteria:

1. Subjects had clinically significant hydronephrosis that could not be relieved by nephrostomy or urethral stenting, as determined by the investigator.
2. Other active malignancies within 2 years prior to the first administration. Subjects with locally curable tumors that appear to be cured, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the breast, were not excluded.
3. Have received other study drugs or study devices within 4 weeks prior to the first administration.
4. Concurrent enrollment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study. (It was defined as more than 4 weeks between the first administration of the drug in the study and the last administration of the drug in the previous clinical study or more than 5 half-lives of the drug in the study)
5. An active infection requiring systemic therapy.
6. Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 1000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <1000 IU/ mL), and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
7. Known history of active tuberculosis (TB),In patients suspected of having active tuberculosis, chest x-rays, sputum, and clinical signs and symptoms should be examined for exclusion.
8. Receipt of live or attenuated vaccination within 30 days prior to the first administration, or plan to receive live or attenuated vaccine during the study.
9. There are any of the following cardiovascular and cerebrovascular diseases or risk factors for cardiovascular and cerebrovascular diseases:

   Myocardial infarction, unstable angina pectoris, pulmonary embolism, acute/persistent myocardial ischemia, cerebrovascular accident, transient ischemic attack, or other arteriovenous thrombosis, embolism, or ischemic events that are clinically significant or require pharmacological intervention occurred within 6 months prior to initial administration.

   Symptomatic congestive heart failure (classified as 3 or 4 according to the New York Heart Association functional classification) occurring within 6 months before the first administration.

   Unstable arrhythmias or degree II/III atrioventricular blocks requiring pharmacological intervention occurred within 6 months prior to initial administration.
10. Known history of serious hypersensitivity reaction to other monoclonal antibodies.
11. Pregnant or lactating women.
12. Any condition that the investigator believes may result in a risk of receiving the study drug or combination therapy, or that would interfere with the evaluation of the study drug or with patient safety or analysis of the study results.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. recurrent or metastatic cervical cancer, not amenable to curative surgery or concurrent chemoradiotherapy, no prior systemic therapy for persistent, recurrent or metastatic disease.
  2. subjects have demonstrated radiologically confirmed disease progression during or after last treatment, subjects will have no more than 2 lines of systemic therapy in the recurrence or metastatic stages.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | from the first drug administration up to two years
  ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | from the first drug administration up to two years
  Disease control rate (DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR and PR and stable disease(SD) per RECIST v1.1.
progression-free survival (PFS) | from the first drug administration up to two years
  Progression-free survival (PFS) is defined as the time from the first dose of investigational products until documentation of PD (as per RECIST v1.1) or death due to any cause, whichever occurs first.
overall survival (OS) | from the first drug administration up to two years
  Overall survival (OS) is defined as the time from the first dose of investigational products until death due to any cause.
Incidence and severity of adverse events(AEs) | from the first drug administration up to two years
  Incidence and severity of AEs is aim to evaluate the safety of Cadonilimab in combination with other treatments.